CLINICAL TRIAL: NCT05042167
Title: The Acute Effect of High-load Resistance Exercise on Inflammation in Young and Older Adults
Brief Title: The Effect of Resistance Exercise on Inflammation in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202012HM020
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Aging; Inflammatory Response
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-load resistance exercise (Experimental): Subjects in high-load trial performed 3 sets per exercise, 8 repetitions with load of 70%-1RM with 90 sec of rest between sets, followed by a fourth set to voluntary failure.
  Interventions: Other: Resistance exercise
- Sedentary control (No Intervention): Subjects in control trial stayed sedentary during the period.

INTERVENTIONS:
Other: Resistance exercise — 4 total resistance exercises that target all major muscle groups.
  Arms: High-load resistance exercise

SUMMARY:
Healthy young and older adults will complete two trials in a randomized crossover counter-balanced order, including resistance exercise and sedentary control. During each trial, blood samples will be collected.

The investigators hypothesized that an acute bout of resistance exercise exert different inflammation responses in young and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80
* Healthy male
* Without experience of resistance training

Exclusion Criteria:

* No acute or chronic musculoskeletal symptoms
* Smoking
* Alcohol or drug abuse
* Fail to conduct resistance exercise

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in biomarkers of inflammation | 24-hour during each study intervention
  Biomarkers of inflammation will be measured such as IL-10 in pg/mL, IL-6 in pg/mL, TNF-α in pg/mL.

SECONDARY OUTCOMES:
Changes in glucose | 24-hour during each study intervention
  glucose in mg/dL
Changes in metabolic parameters | 24-hour during each study intervention
  Metabolic parameters will be measured such as TC in mg/dL, TG in mg/dL, and HDL in mg/dL.
Changes in biomarkers of muscle damage | 24-hour during each study intervention
  Biomarkers of muscle damage will be measured such as CK in U/L and LDH in U/L.
Changes in molecular markers in peripheral blood mononuclear cells (PBMC) | 24-hour during each study intervention
  Molecular markers in PBMC will be measured such as STAT3 in arbitrary units, IKK in arbitrary units, IkB in arbitrary units, p65 in arbitrary units, SOCS3 in arbitrary units, AMPK in arbitrary units, and SIRT1 in arbitrary units.
Changes in complete blood count (CBC) | 24-hour during each study intervention
  The white blood cell count and the count of each white blood cell type will be measured.
Borgs Ratings of Perceived Exertion (RPE) | 1-hour during each exercise intervention
  Borgs RPE is a method of estimating exertion rating, based on a 6 to 20 rating scale (6 being the no exertion at all, 20 being maximal exertion).

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wen Liu, Ph.D., Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai SH, Cheng HC, Little JP, Islam H, Liu HW. Elevated Plasma IL-6 Coincides with Activation of STAT3 in PBMC After Acute Resistance Exercise. Med Sci Sports Exerc. 2024 Nov 1;56(11):2117-2124. doi: 10.1249/MSS.0000000000003503. PMID 39475859